CLINICAL TRIAL: NCT07311967
Title: Short-Term Health Outcomes of Cooking UFP Exposure
Acronym: UFP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Illinois Chicago, Chicago, Illinois (Unknown)
Responsible Party: Principal Investigator, Mehdi Amouei Torkmahalleh, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY2025-1120
Record Dates: First submitted 2025-11-28; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Function Decline; Air Pollution Exposure; Respiratory Inflammation
Keywords: Cooking emissions; Neurocognitive function; Respiratory symptoms; Ultrafine particles
MeSH Terms: conditions — Signs and Symptoms, Respiratory | interventions — Gases

STUDY DESIGN:
Intervention Model Description: This study uses a two-period randomized crossover design in which each participant completes both conditions: a control session with clean indoor air and an exposure session involving cooking-generated ultrafine particles. The two sessions occur on consecutive days in the same controlled exposure chamber, and participants serve as their own control to allow within-subject comparisons of respiratory and cognitive responses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (Clean Indoor Air) (Other): Participants will complete a control study session conducted in a controlled exposure chamber with clean indoor air and no cooking activity. Respiratory, cognitive, and physiological outcomes will be assessed during the session.
  Interventions: Other: Clean Indoor Air Exposure (Control)
- Cooking Emissions Exposure (Experimental): Participants will complete an exposure study session conducted in the same controlled exposure chamber during which cooking activities generate ultrafine particles. Respiratory, cognitive, and physiological outcomes will be assessed during the session.
  Interventions: Other: Exposure to Cooking-Generated Ultrafine Particles and Gases

INTERVENTIONS:
Other: Clean Indoor Air Exposure (Control) — Participants will be exposed to clean indoor air in a controlled exposure chamber with no cooking activity. This condition serves as the control session for within-subject comparisons.
  Arms: Control Condition (Clean Indoor Air)
Other: Exposure to Cooking-Generated Ultrafine Particles and Gases — Participants will be exposed to cooking-generated ultrafine particles and associated gases in a controlled exposure chamber during standardized cooking activities.
  Arms: Cooking Emissions Exposure

SUMMARY:
This study examines the short-term respiratory and cognitive effects of exposure to ultrafine particles (UFPs) generated during typical household cooking. Healthy adults will complete two 6-hour sessions in a controlled exposure chamber at the University of Illinois Chicago: one control day with clean indoor air and one exposure day during which standardized cooking (frying potatoes and grilling beef) is performed by research staff. Participants will not cook or handle food. Lung function will be measured using peak expiratory flow (PEF), and cognitive performance will be assessed using validated tests including the Hopkins Verbal Learning Test-Revised and the Processing Speed Index from the WAIS-IV. Airborne particle and gas concentrations in the chamber will be continuously monitored to ensure that exposures remain within levels typical of everyday home cooking. Findings will help characterize acute physiological responses to indoor cooking emissions and inform future research on indoor air quality and potential mitigation strategies.

DETAILED DESCRIPTION:
This study evaluates the short-term respiratory and cognitive responses to controlled exposure to cooking-generated ultrafine particles (UFPs). Cooking emissions are one of the most common sources of indoor particulate pollution, yet their acute physiological effects remain poorly characterized. To address this gap, the study uses a controlled exposure chamber environment that reproduces typical household cooking conditions while allowing precise measurement of airborne particle and gas concentrations.

Healthy adult volunteers will participate in two study sessions conducted on consecutive days. On the exposure day, research staff will prepare a standardized meal (frying potatoes and grilling beef) inside the chamber to generate UFPs and co-emitted gases at levels representative of home cooking. On the control day, participants remain in the same chamber but without any cooking activity. Participants will spend approximately six hours in the chamber each day and will remain at rest except during scheduled assessments.

The study employs a randomized two-period crossover design so each participant serves as their own control. Lung function and cognitive performance are assessed multiple times on each day using validated instruments. Air quality is monitored continuously using particle sizing instruments, particle mass monitors, and a gas analyzer to characterize exposure conditions. Pre-defined stopping rules and ventilation procedures are implemented if concentrations exceed levels typical of household cooking.

This study is designed to generate preliminary U.S.-based data on the immediate effects of cooking-related UFP exposure on respiratory function and cognitive performance. Findings will help define exposure-response patterns, support future NIH and American Lung Association proposals, and improve understanding of indoor air quality impacts in everyday environments.

ELIGIBILITY:
Inclusion Criteria

Adults 18 years of age or older

Able to understand and speak English sufficiently to complete cognitive testing

Able and willing to complete two consecutive study sessions lasting approximately 6 hours each

Able to avoid cooking, toasting, and fume-generating household activities (e.g., strong cleaning products, ironing, hair drying) for 24 hours before each session

Able to avoid tobacco, marijuana, vaping, and alcohol use as specified in the study protocol

Able to provide informed consent

Exclusion Criteria

Younger than 18 years old

Pregnant or planning pregnancy during study participation

Current smoking or use of:

Cigarettes

E-cigarettes or vaping devices

Marijuana

Shisha/hookah

Binge drinking, heavy alcohol use, or inability to abstain from alcohol for 24 hours before study visits

Restaurant chefs or individuals who perform frequent commercial-level cooking

Individuals who cook two or more frying or grilling meals per day at home

Cooking anxiety or mageirocophobia

Any diagnosed neurological disease, including stroke, seizure disorder, multiple sclerosis, traumatic brain injury, dementia, or similar conditions

Any significant respiratory disease, including:

Chronic obstructive pulmonary disease (COPD)

Untreated severe asthma

Chronic bronchitis or other major lung disease

Any significant psychiatric condition, including:

Schizophrenia spectrum disorder

Untreated substance use disorder

Severe mood disorder

Severe anxiety disorder

Claustrophobia or anxiety in enclosed spaces (if severe enough to interfere with chamber procedures)

Inability to comply with study procedures or safety requirements

Any medical or psychological condition that, in the judgement of the investigators, may increase risk or interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hopkins Verbal Learning Test-Revised (HVLT-R) Total Recall Score | Measured at baseline and at approximately 1, 2, 3, and 5 hours after session start on both study days
  Cognitive performance related to verbal memory will be assessed using the Hopkins Verbal Learning Test-Revised (HVLT-R). The primary metric will be the change in HVLT-R Total Recall Score between exposure and control conditions, calculated from repeated assessments to evaluate short-term cognitive effects of ultrafine particle exposure.
Change in Peak Expiratory Flow (PEF) | Measured at baseline and at approximately 1, 2, 3, and 5 hours after session start on both study days
  Peak Expiratory Flow (PEF) will be measured using a handheld peak flow meter to assess short-term changes in lung function following exposure to cooking-generated ultrafine particles compared with the clean-air control day. Changes are evaluated within subjects using repeated measurements across both conditions.
Change in WAIS Symbol Search Raw Score | Measured at baseline and at approximately 1, 2, 3, and 5 hours after session start on both study days
  Cognitive performance related to processing speed and visual attention will be assessed using the Symbol Search subtest of the Wechsler Adult Intelligence Scale (WAIS). The primary metric will be the change in WAIS Symbol Search raw score between exposure and control conditions, calculated from repeated assessments to evaluate short-term cognitive effects of ultrafine particle exposure.

SECONDARY OUTCOMES:
Ultrafine Particle Number Size Distribution in particles/cm3 | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods.
  Ultrafine particle number size distributions will be measured using a Scanning Mobility Particle Sizer (SMPS) and Partector 2 Pro. These measurements characterize exposure conditions and allow correlation with physiological responses.
Fine Particle Mass Concentrations (PM2.5) in microgram/cm3 | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods
  Particle mass concentrations (PM2.5) will be measured using a DustTrak DRX monitor to quantify particulate exposure profiles during cooking and control sessions. These measurements characterize exposure conditions and allow correlation with physiological responses.
Total Volatile Organic Compound (VOC) concentration in ppm | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods
  Concentrations of over 50 volatile organic compounds (VOCs) will be monitored using FTIR spectroscopy (Gasmet DX4040) to characterize exposure to total VOC concentration during cooking. The concentration of individual gases will be add up to quantify total VOC concentration.
CO2 concentration in ppm | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods
  Description: Concentrations of CO2 will be monitored using Atmocube, Atmo, USA instrument. This measurement characterize exposure conditions and allow correlation with physiological responses.
CO concentration in ppm | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods
  Description: Concentrations of CO will be monitored using FTIR spectroscopy (Gasmet DX4040) to characterize exposure to CO during cooking. The
NO2 concentration in ppm | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods
  Concentrations of NO2 will be monitored using FTIR spectroscopy (Gasmet DX4040) to characterize exposure to NO2 during cooking.

OTHER OUTCOMES:
Temperature Condition in Exposure Chamber | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods
  Ambient temperature will be recorded to ensure environmental conditions remain consistent and to support interpretation of particle behavior.
Number of Participants Reporting Acute Symptoms During Study Sessions | Assessed at baseline and at approximately 1, 2, 3, and 5 hours after session start on control and exposure days
  Participant-reported symptoms related to tolerability of the study procedures and exposure will be assessed using a standardized symptom checklist administered by study staff. Symptoms assessed will include throat or eye irritation, cough, headache, dizziness, and nausea. The outcome measure will be the number of participants reporting one or more symptoms during each study session.
Relative Humidity Condition in Exposure Chamber | Continuously measured average concentration with one minute intervals during each study session on control and exposure days, from session start to session end (approximately 5 hours per session), across both study periods
  Relative Humidity in the chamber will be recorded to ensure environmental conditions remain consistent and to support interpretation of particle behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Amouei Torkmahalleh, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- UIC, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study does not collect biospecimens and all data are used solely for the analyses specified in the protocol. Data are stored in coded form and are not intended for secondary research use. In addition, screening data for ineligible individuals are destroyed within 3 days, and no identifiable information is retained beyond what is required for regulatory documentation. Only aggregate, de-identified results may be shared with participants upon request, but individual-level datasets will not be made available to external researchers.

REFERENCES:
- Available data/document: Study Protocol — https://uofi.box.com/s/3vs1mzdcyzsbafojrytxk3d1n6ed45z8
- Available data/document: Informed Consent Form — https://uofi.box.com/s/5g14s3norggukhl3oyrh6vy6mm8f1vpp
- Available data/document: Recruitment Email — https://uofi.box.com/s/sr3cztrcr8av6ydub4s76kxo7co5slck
- Available data/document: Screening Materials — https://uofi.box.com/s/0ixpcy9goxx5ggguo8vurdb6ncq3lne7